CLINICAL TRIAL: NCT06347783
Title: The Effect of Automated Insulin Delivery on Sleep Compared to Multiple Daily Injections in Pediatric Patients With Type 1 Diabetes
Brief Title: Automated Insulin Delivery vs. Injections: Sleep Impact in Pediatric Type 1 Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Rachel Palting, Pediatric endocrinology fellow, Oregon Health and Science University
Other Study IDs: STUDY00026893
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Insulin Infusion Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Child/parent dyad: Study group will consist of 40 participant dyads - a pediatric patient with type 1 diabetes and one of their caregivers. At the beginning of the study, the patient's treatment should consist of multiple daily insulin injections and a continuous glucose monitor, and during this time, sleep will be evaluated through a FitBit and surveys. Then patient will be started on an insulin pump of their choice (Omnipod 5, Tandem, etc), and sleep will be re-evaluated 1-2 months after pump initiation.
  Interventions: Device: Insulin pump

INTERVENTIONS:
Device: Insulin pump — Continuous subcutaneous insulin therapy.

SUMMARY:
The purpose of the study is to learn about the effect of insulin pumps on sleep in pediatric patients with type 1 diabetes and their caregivers. We are hoping to find out if insulin pumps improve sleep, worsen sleep, or have no effect at all. We are hoping to also explore the relationship between insulin pumps, sleep, and overnight blood sugar control. Your information will not be stored and used for future research.

The goal of this observational study is learn about the effect of insulin pumps on sleep in pediatric patients with type 1 diabetes and their caregivers. The main questions it aims to answer are:

Do insulin pumps improve sleep, worsen sleep or have no effect at all? What is the relationship between insulin pumps, sleep, and overnight blood sugar control?

Participants will be asked to:

* Complete questionnaires regarding demographic data and diabetes history.
* Complete surveys regarding sleep quality before and after starting an insulin pump.
* Wear a FitBit during sleep for 2 weeks and fill out daily sleep diaries over a 2 week period prior to starting an insulin pump.

After 1-2 months after initiation of an insulin pump, participants will be asked again to:

* Complete surveys regarding sleep quality
* Wear a FitBit during sleep for 2 weeks
* Fill out daily sleep diaries over the same 2 week period.

ELIGIBILITY:
Inclusion Criteria:

i. Diagnosis: Type 1 diabetes for at least 6 months ii. Age: Participants must be aged between 6-18 years at time of enrollment iii. Treatment modality: Participants must be currently receiving treatment for Type 1 Diabetes through multiple daily injections of insulin, with concomitant use of a continuous glucose monitor, with data sharing through Clarity. Participants must be eligible for an insulin pump, based on individual provider discretion.

iv. Smartphone access, ability to download FitBit application. v. Language: Participants and their guardians must be able to understand and communicate in the primary language(s) used for study-related instructions and questionnaires, which include a demographic survey, questions about diabetes history, two surveys regarding patient and caregiver sleep, and a daily sleep diary.

vi. Informed Consent: Participants (if aged 18 or older) or their legal guardians must provide informed consent for participation in the study.

Exclusion Criteria:

i. Diagnosis: Participants with a diagnosis other than Type 1 Diabetes (e.g. Type 2 Diabetes or MODY).

ii. Age: Participants outside the age range of 6 to 18 years. iii. Treatment modality:

1. Participants currently not receiving multiple daily injections of insulin.
2. Participants currently not using a continuous glucose monitor. iv. Participants ineligible for an insulin pump. v. No access to smartphone vi. Inadequate language proficiency: Participants or guardians that cannot communicate effectively in the primary study language.

vii. If a participant is otherwise eligible for the study, a modification may be submitted to the IRB to include the participant in the study. However, language barrier is not an obstacle for a patient to receive standard care in the clinic.

viii. Pregnancy: Pregnancy can significantly affect insulin requirements and sleep patterns.

ix. Allergy or Sensitivity: Participants with known allergies or sensitivities to materials used in Fitbit devices or related equipment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include pediatric patients diagnosed with Type 1 Diabetes ages 6-18 years currently using multiple daily injections combined with a continuous glucose monitor, eligible for an insulin pump. For this pilot study, a sample size of 40 patients with their caregivers, for a total of 80 individuals.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Sleep duration | 4 months
  Number of hours and minutes measured by FitBit
Sleep efficiency | 4 months
  The percentage of time spent asleep while in bed, calculated as the ratio of total sleep time to total time spent in bed.

SECONDARY OUTCOMES:
Sleep Disturbance Scale for Children | 4 months
  Measures sleep disturbances in children and adolescents, with a T-score ranging from 38 to >100
Promis Short Form 8a | 4 months
  Assess sleep disturbances in caregivers, converts a raw score (8-40) to a T-score (30.5-77.5).

OTHER OUTCOMES:
Time in range | 4 months
  Measures of blood glucose levels during sleep, frequency of hypoglycemic/hyperglycemic events obtained through CGM data.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Palting, DO, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaser SS, Bergner EM, Hamburger ER, Bhatia S, Lyttle M, Bell GE, Slaughter JC, Malow BA, Simmons JH. Pilot Trial of a Sleep-Promoting Intervention for Children With Type 1 Diabetes. J Pediatr Psychol. 2021 Mar 18;46(3):304-313. doi: 10.1093/jpepsy/jsaa105. PMID 33180913
- [Background] Reutrakul S, Thakkinstian A, Anothaisintawee T, Chontong S, Borel AL, Perfect MM, Janovsky CC, Kessler R, Schultes B, Harsch IA, van Dijk M, Bouhassira D, Matejko B, Lipton RB, Suwannalai P, Chirakalwasan N, Schober AK, Knutson KL. Sleep characteristics in type 1 diabetes and associations with glycemic control: systematic review and meta-analysis. Sleep Med. 2016 Jul;23:26-45. doi: 10.1016/j.sleep.2016.03.019. Epub 2016 Jun 8. PMID 27692274
- [Background] Leese GP, Wang J, Broomhall J, Kelly P, Marsden A, Morrison W, Frier BM, Morris AD; DARTS/MEMO Collaboration. Frequency of severe hypoglycemia requiring emergency treatment in type 1 and type 2 diabetes: a population-based study of health service resource use. Diabetes Care. 2003 Apr;26(4):1176-80. doi: 10.2337/diacare.26.4.1176. PMID 12663593
- [Background] Jaser SS, Foster NC, Nelson BA, Kittelsrud JM, DiMeglio LA, Quinn M, Willi SM, Simmons JH; T1D Exchange Clinic Network. Sleep in children with type 1 diabetes and their parents in the T1D Exchange. Sleep Med. 2017 Nov;39:108-115. doi: 10.1016/j.sleep.2017.07.005. Epub 2017 Jul 18. PMID 29157581
- [Background] Matyka KA, Crawford C, Wiggs L, Dunger DB, Stores G. Alterations in sleep physiology in young children with insulin-dependent diabetes mellitus: relationship to nocturnal hypoglycemia. J Pediatr. 2000 Aug;137(2):233-8. doi: 10.1067/mpd.2000.107186. PMID 10931417
- [Background] Brod M, Pohlman B, Wolden M, Christensen T. Non-severe nocturnal hypoglycemic events: experience and impacts on patient functioning and well-being. Qual Life Res. 2013 Jun;22(5):997-1004. doi: 10.1007/s11136-012-0234-3. Epub 2012 Jul 24. PMID 22825805
- [Background] O'Reilly M, O'Sullivan EP, Davenport C, Smith D. "Dead in bed": a tragic complication of type 1 diabetes mellitus. Ir J Med Sci. 2010 Dec;179(4):585-7. doi: 10.1007/s11845-010-0519-x. Epub 2010 Jul 24. PMID 20658206
- [Background] McDonough RJ, Clements MA, DeLurgio SA, Patton SR. Sleep duration and its impact on adherence in adolescents with type 1 diabetes mellitus. Pediatr Diabetes. 2017 Jun;18(4):262-270. doi: 10.1111/pedi.12381. Epub 2016 Mar 30. PMID 27028035
- [Background] Jaser SS, Ellis D. Sleep in Adolescents and Young Adults with Type 1 Diabetes: Associations with Diabetes Management and Glycemic Control. Health Psychol Behav Med. 2016 Jan 1;4(1):49-55. doi: 10.1080/21642850.2015.1135293. Epub 2016 Mar 2. PMID 27081578
- [Background] Monzon A, McDonough R, Meltzer LJ, Patton SR. Sleep and type 1 diabetes in children and adolescents: Proposed theoretical model and clinical implications. Pediatr Diabetes. 2019 Feb;20(1):78-85. doi: 10.1111/pedi.12797. Epub 2018 Dec 4. PMID 30447038
- [Background] Goel N, Rao H, Durmer JS, Dinges DF. Neurocognitive consequences of sleep deprivation. Semin Neurol. 2009 Sep;29(4):320-39. doi: 10.1055/s-0029-1237117. Epub 2009 Sep 9. PMID 19742409
- [Background] Quist JS, Sjodin A, Chaput JP, Hjorth MF. Sleep and cardiometabolic risk in children and adolescents. Sleep Med Rev. 2016 Oct;29:76-100. doi: 10.1016/j.smrv.2015.09.001. Epub 2015 Sep 12. PMID 26683701
- [Background] Dahl RE, Lewin DS. Pathways to adolescent health sleep regulation and behavior. J Adolesc Health. 2002 Dec;31(6 Suppl):175-84. doi: 10.1016/s1054-139x(02)00506-2. PMID 12470913